CLINICAL TRIAL: NCT06832839
Title: Study on the Mechanism of Cognitive Impairment in Patients with Moyamoya Disease
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2024-112-02
Record Dates: First submitted 2025-01-26; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Moyamoya Disease
Keywords: Cognitive Impairment; Moyamoya Disease
MeSH Terms: conditions — Moyamoya Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Revascularization — Revascularization

SUMMARY:
The purpose of this study is to comprehensively evaluate the risk factors for cognitive decline in patients with moyamoya disease, identify imaging target areas associated with cognitive damage in the brain, and explore the changes in brain structure and functional networks resulting from cerebral revascularization, as well as their relationship with cognitive improvement.

DETAILED DESCRIPTION:
Moyamoya disease (MMD) is a chronic occlusive-stenosis cerebrovascular disease that characterized by the stenosis of internal carotid artery termination and the formation of net-like vessel. It is a multifactorial disease caused by genetic, inflammatory, immunological and other environmental factors. The specific pathogenesis of MMD is still unclear. The treatment modalities of revascularization and conservative management have been used in patients with MMD. Due to the long-term low perfusion state of brain tissue, most patients with MMD experience varying degrees of cognitive dysfunction, although the underlying mechanisms remain unclear. We will employ a combination of 256-lead high-density electroencephalography, multimodal magnetic resonance imaging, and biological samples to conduct a comprehensive evaluation of the risk factors associated with cognitive decline in patients with MMD. Our objectives include identifying target imaging areas indicative of cognitive damage in the brain and exploring the structural and functional changes in the cerebral network resulting from revascularization, as well as their relationship with cognitive improvement.

ELIGIBILITY:
Inclusion Criteria:

* The admission cerebral angiography (DSA) examination fulfills the diagnostic criteria for moyamoya disease.
* Please sign the informed consent form.
* Participants must be between 18 and 60 years of age.

Exclusion Criteria:

* Patients with concurrent atherosclerosis, autoimmune diseases, meningitis, brain tumors, Down syndrome, craniocerebral trauma, prior radioactive head irradiation, or hyperthyroidism, which may result in secondary cerebrovascular lesions leading to symptoms associated with smoke syndrome.
* Individuals younger than 18 years or older than 60 years.
* Those with contraindications for magnetic resonance imaging.
* Patients who are unable to complete cognitive brain assessments

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Consecutive patients diagnosed with MMD in Beijing Tiantan Hospital will be recruited. Eligibility will be determined through a checklist of inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in composite score of neurocognitive function at 6 months after treatment. | 6 months during follow-up
  The composite score of neurocognitive function, including Weschsler Adult Intelligence Scale-4th Edition (WAIS-IV), MATRICS Consensus Cognitive Battery (MCCB), Montreal Cognitive Assessment (MoCA), Auditory Verbal Learning Test (AVLT), Rey-Osterrieth complex figure (ROCF), Trail Making Test (TMT), Stroop test, Verbal Fluency Test (VFT), and Boston Naming Test (BNT) will be collected before and 6 months after treatment.

SECONDARY OUTCOMES:
Changes in composite score of neurocognitive function at 12 and 24 months after treatment. | 12 and 24 months during follow-up
  The composite score of neurocognitive function, including Weschsler Adult Intelligence Scale-4th Edition (WAIS-IV), MATRICS Consensus Cognitive Battery (MCCB), Montreal Cognitive Assessment (MoCA), Auditory Verbal Learning Test (AVLT), Rey-Osterrieth complex figure (ROCF), Trail Making Test (TMT), Stroop test, Verbal Fluency Test (VFT), and Boston Naming Test (BNT) will be collected before and 12 and 24 months after treatment.
Rate of participants experiencing cerebrovascular events (TIA, infarction and hemorrhage) within 6, 12 and 24 months after treatment. | 6, 12 and 24 months during follow-up
Changes in neurological function assessed by modified Rankin scale (mRS) at 6, 12, and 24 months following treatment. | 6, 12 and 24 months during follow-up
Changes in neurological function assessed by National Institute of Health stroke scale (NIHSS) at 6, 12, and 24 months following treatment. | 6, 12 and 24 months during follow-up
Changes in cerebral blood perfusion assessed by arterial spin labeling (ASL) at 6, 12, and 24 months after treatment. | 6, 12 and 24 months during follow-up
Hemodynamic changes at the terminal segment of internal carotid artery assessed by computational fluid dynamics (CFD) at 6, 12, and 24 months after treatment. | 6, 12 and 24 months during follow-up
Morphological changes at the terminal segment of internal carotid artery and middle cerebral artery wall assessed by high-resolution vessel wall imaging at 6, 12, and 24 months after treatment. | 6, 12 and 24 months during follow-up
Changes in Power Spectral Density (PSD) assessed by electroencephalography (EEG) at 6, 12, and 24 months after treatment will be measured. | 6, 12 and 24 months during follow-up
Changes in Phase Locking Value (PLV) assessed by electroencephalogram (EEG) at 6, 12, and 24 months after treatment will be measured. | 6, 12 and 24 months during follow-up
Changes in Phase-Lag Index (PLI) assessed by electroencephalogram (EEG) at 6, 12, and 24 months after treatment will be measured. | 6, 12 and 24 months during follow-up
Changes in Degree Centrality assessed by multimodal MRI at 6, 12, and 24 months after treatment. | 6, 12 and 24 months during follow-up
Changes in Clustering Coefficient assessed by multimodal MRI at 6, 12, and 24 months after treatment. | 6, 12 and 24 months during follow-up
Changes in Structural Connectivity Strength assessed by multimodal MRI at 6, 12, and 24 months after treatment. | 6, 12 and 24 months during follow-up
Changes in Network Density assessed by multimodal MRI at 6, 12, and 24 months after treatment. | 6, 12 and 24 months during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China, China